CLINICAL TRIAL: NCT05104554
Title: School-Based Assessment of Micronutrient Interventions in Adolescents (SAMIA) in Zanzibar
Acronym: SAMIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Africa Academy for Public Health (Other); Zanzibar Association of People Living with HIV/AIDS (ZAPHA+) (Unknown)
Responsible Party: Principal Investigator, Wafaie Fawzi, Professor of Nutrition, Epidemiology, and Global Health, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB20-1108-2
Record Dates: First submitted 2021-10-21; First posted 2021-11-03 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Anemia
Keywords: Anemia; Multiple Micronutrient Supplementation (MMS); Iron and Folic Acid (IFA); Nutrition; Adolescent Health
MeSH Terms: conditions — Anemia | interventions — Iron; Folic Acid

STUDY DESIGN:
Intervention Model Description: Schools will be randomly assigned to weekly iron and folic acid (IFA) supplementation, daily multiple micronutrient supplements (MMS), or control. Supplementation will be conducted continuously over the course of the first year. Baseline and end-line surveys will be conducted to collect demographic information and assess outcomes. In the second year of the study, the more effective supplementation strategy (IFA or MMS) will be scaled up to all study schools and the outcomes will be re-assessed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Weekly IFA (Experimental): Receive weekly IFA
  Interventions: Dietary Supplement: Iron and folic acid (IFA)
- Daily MMS (Experimental): Receive daily MMS (including iron and folic acid as components)
  Interventions: Dietary Supplement: Multiple Micronutrient Supplement (MMS)
- Control (No Intervention)

INTERVENTIONS:
Dietary Supplement: Iron and folic acid (IFA) — IFA: Weekly regimen of one tablet containing iron (60 mg) and folic acid (2800 μg)
  Arms: Weekly IFA
Dietary Supplement: Multiple Micronutrient Supplement (MMS) — MMS: Daily regimen of one multiple micronutrient tablet containing fifteen micronutrients in the United Nations International Multiple Micronutrient Preparation (UNIMMAP) preparation. Composition includes vitamin A (800 ug), vitamin D (5 ug), vitamin E (10 mg), vitamin C (70 mg), vitamin B1 (1.4 mg), vitamin B2 (1.4 mg), niacin (18 mg), vitamin B6 (1.9 mg), vitamin B12 (2.6 ug), folic acid (400 ug), iron (30 mg), zinc (15 mg), copper (2 mg), selenium (65 ug), and iodine (150 ug).
  Arms: Daily MMS

SUMMARY:
This purpose of this study is to assess effects of iron and folic acid supplementation and multiple micronutrient supplementation on anemia status and school performance/attendance among in-school adolescents in Zanzibar, Tanzania.

DETAILED DESCRIPTION:
This study aims to implement and evaluate micronutrient supplementation interventions to improve adolescent nutrition, health and education in Zanzibar. Findings from this study will clarify the optimal supplementation strategy (iron and folic acid alone or adding other essential nutrients) and provide a basis for scale up of national micronutrient supplementation programs to benefit the adolescent population as a whole in Zanzibar.

This will be a cluster randomized study with 3 arms. At the beginning of the academic year, 42 schools will be enrolled (14 schools per arm) to receive either 1) supplementation with weekly iron and folic acid (IFA); 2) supplementation with daily multiple micronutrient supplements (MMS) (including iron and folic acid as components); or 3) to serve as controls. Students in intervention schools will receive supplementation and students in control schools will receive the usual care (which does not include supplementation but does include existing curriculum on nutrition and water, sanitation and hygiene [WASH]). The program will be evaluated at the end of year 1, comparing effects of weekly IFA and daily MMS on anemia status and school attendance/performance. The more effective strategy (MMS or IFA) will be scaled up to all the study schools for year 2 of the intervention, and the outcomes will be re-assessed.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 10-17 years
* Enrolled in secondary school form 1 at study initiation
* Member of one of the selected classes in a participating school
* Consent provided by the parent
* Assent provided by the adolescent
* Fluency in Swahili and/or English

Exclusion Criteria:

* No informed consent from parent or assent from adolescent
* Self-reported pregnancy

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2480 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Anemia status | Up to one year
  Anemia will be defined based on the sex- and age- specific WHO cutoffs:
  1. Children 12-14 years: < 120 g/L
  2. Non-pregnant women ≥ 15 years: < 120 g/L
  3. Pregnant women: < 110 g/L
  4. Men ≥ 15 years: < 130 g/L

SECONDARY OUTCOMES:
School attendance | Up to one year
  Number of days of missed school per student
School retention | Up to one year
  Number of students who drop out of school
School performance | Up to one year
  Percent of students who pass to the next grade at the end of the year

CONTACTS AND LOCATIONS:
Overall Officials: Wafaie W Fawzi, MBBS, MPH, MS, DrPH, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- Zanzibar Association for People Living with HIV/AIDS, Welezo, Zanzibar, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yusufu I, Cliffer IR, Yussuf MH, Anthony C, Mapendo F, Abdulla S, Masanja M, Tinkasimile A, Ali AS, Mwanyika-Sando M, Fawzi W. Factors associated with anemia among school-going adolescents aged 10-17 years in Zanzibar, Tanzania: a cross sectional study. BMC Public Health. 2023 Sep 18;23(1):1814. doi: 10.1186/s12889-023-16611-w. PMID 37723498
- [Derived] Cliffer IR, Yussuf MH, Millogo O, Mwanyika-Sando M, Barry Y, Yusufu IS, Hemler EC, Sie A, Tinkasimile A, Compaore G, Ali AS, Kouanda I, Wang D, Mosha D, Fawzi W. Scaling-up high-impact micronutrient supplementation interventions to improve adolescents' nutrition and health in Burkina Faso and Tanzania: protocol for a cluster-randomised controlled trial. BMJ Open. 2023 Feb 15;13(2):e063686. doi: 10.1136/bmjopen-2022-063686. PMID 36792333